CLINICAL TRIAL: NCT07297394
Title: Mechanisms of Maternal Immune Tolerance in Early Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-02262;bb25GobrechtKeller
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy; Immune Tolerance; In Vitro Fertilization
Keywords: Maternal Immune Tolerance; Early Pregnancy; Immune Regulation; T cells; Cytokines
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing IVF and early pregnancy: This cohort includes women undergoing in vitro fertilization (IVF)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood samples will be analyzed before and during early pregnancy as well as after early miscarriage

SUMMARY:
This study explores the mechanisms of maternal immune tolerance in early pregnancy by characterizing immune cell profiles and functional pathways during the first trimester. The goal is to identify immunological factors that support healthy gestation and prevent complications such as miscarriages.

DETAILED DESCRIPTION:
Maternal immune tolerance is essential for a successful pregnancy, as the maternal immune system must accept the semi-allogeneic fetus while maintaining defense against pathogens. Failure in this delicate balance can lead to complications such as recurrent miscarriage, preeclampsia, or implantation failure. Although several immune cell types, including T cells and regulatory pathways, are thought to play a role, the precise mechanisms underlying maternal immune adaptation during early pregnancy remain poorly understood.

This observational study investigates immunological changes occurring before and during early pregnancy and miscarriage in women undergoing in vitro fertilization (IVF). Blood samples will be collected at multiple predefined time points: prior to embryo transfer and during the first trimester of pregnancy as well as after miscarriage. These samples will be analyzed for immune cell composition, activation status, and cytokine profiles using advanced immunological assays. The longitudinal design allows for tracking dynamic changes in immune regulation from pre-implantation through early gestation.

The primary objective is to identify cellular and molecular signatures associated with maternal immune tolerance and successful implantation. Insights gained from this study may inform future strategies to predict and prevent pregnancy complications such as early miscarriage related to immune dysregulation.

ELIGIBILITY:
Inclusion Criteria:

Blood from patients will be included before and during pregnancies (or failed implantation) conceived through IVF/ICSI (Intracytoplasmic Sperm Injection) treatment and in case of miscarriage.

1. where the patient (pregnant person) was ≥ 18 years of age.
2. where the patient (pregnant person) signed a written informed consent.

Exclusion Criteria:

1. Certain maternal infections (HIV, Hepatitis B, Hepatitis C, Syphilis)
2. Patients under immunosuppressive medications (at time of blood sample collection)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing in vitro fertilization (IVF) treatment at the University Hospital Basel who consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Immune cell composition in peripheral blood | Before conception, week 6-7 of pregnancy, and following implantation failure or spontaneous miscarriage, up to 12 weeks of gestation
  Characterization of immune cell subsets (e.g., T cells, regulatory T cells, natural killer cells (NK cells)) in blood samples collected at predefined time points (before embryo transfer and during early pregnancy and in case of early miscarriage).

SECONDARY OUTCOMES:
Transcriptional profiles of peripheral blood mononuclear cell (PBMC) subsets associated with pregnancy outcome (scRNA-seq) | Before conception, week 6-7 of pregnancy, and following implantation failure or spontaneous miscarriage, up to 12 weeks of gestation
  Single-cell RNA sequencing analysis to characterize transcriptional phenotypes of PBMCs. This includes identification of differentially expressed genes, gene modules, and transcription factor activity profiles associated with pregnancy and pregnancy failure.
T-cell and B-cell receptor repertoire dynamics (TCR/BCR sequencing) | Before conception, week 6-7 of pregnancy, and following implantation failure or spontaneous miscarriage, up to 12 weeks of gestation
  Assessment of clonal expansion and contraction in TCR and BCR (B cell receptor) repertoires using bulk and single-cell sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Gobrecht-Keller, MD, Study Director — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No